CLINICAL TRIAL: NCT03297905
Title: Determinants of the Optimal Dose and Sequence of Functional Restoration and Integrative Therapies in Service Members With Neuromusculoskeletal Injury
Brief Title: Functional Restoration and Integrative Therapies in Service Members With Neuromusculoskeletal Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ardith Doorenbos, Professor, University of Washington
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004220
Record Dates: First submitted 2017-08-08; First posted 2017-09-29 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Military
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial (SMART)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complementary and Integrative Therapies (Experimental): Chiropractic, Acupuncture, Yoga, Biofeedback (if indicated), and Foam roller instruction
  Interventions: Behavioral: Complementary and Integrative Therapies
- Standard Rehabilitative Care (Active Comparator): Cognitive Behavioral Therapy (CBT) 60-minute orientation, CBT psychoeducation group, and Physical therapy/occupational therapy
  Interventions: Behavioral: Standard Rehabilitative Care

INTERVENTIONS:
Behavioral: Complementary and Integrative Therapies — Intervention time period is 3 - 6 weeks.
  Arms: Complementary and Integrative Therapies
Behavioral: Standard Rehabilitative Care — Intervention time period is 3 - 6 weeks.
  Arms: Standard Rehabilitative Care

SUMMARY:
This study will (1) compare the effectiveness of standard rehabilitative pain care with complementary and integrative pain therapies; (2) identify subgroups of patients who do and do not respond to the intervention(s); (3) determine the most effective sequencing of the interventions; and (4) determine factors associated with treatment response that can be implemented to support clinical decision-making.

DETAILED DESCRIPTION:
Objectives and Rationale. Pain due to neuromusculoskeletal injuries is a leading cause of disability among active duty military Service members. The injury rate is significant with 628 neuromusculoskeletal injuries per 1000 person-years among active duty military Service members. Neuromusculoskeletal injuries include amputations following battlefield trauma, repetitive motion injuries related to equipment use or weight-bearing postures, and even injuries or strains incurred during off-duty pursuits. Regardless of cause, the effects on both individual Service members and military readiness are significant: Only 13% of Service members being treated primarily for pain ever return to the field.

The Department of Defense (DoD) has recently expanded its capacity to provide both functional restoration (FR) and complementary and integrative medicine (CIM) therapies for neuromusculoskeletal injury, pain, and disability. The proposed research aims to determine the most effective treatment combination, sequence, and duration of standard rehabilitative care (SRC), such as physical and occupational therapy in combination with cognitive behavioral therapy and CIM therapies, such as acupuncture and chiropractic, for Service members preparing to enroll in an intensive FR program that is currently the DoD-recommended treatment. In addition, this study aims to identify ways to predict in advance which patients will respond best to which therapeutic regimens.

Potential Impact. This research has the potential to determine which patients are most likely to benefit from the non-medication pain therapies currently available in all Army Interdisciplinary Pain Management Centers (IPMC) and how these therapies can most effectively be combined to achieve the greatest improvements in pain impact, quality of life and ability to return to duty following injury.

Patients Who Will Benefit. This study will involve active duty Service members referred to an Army IPMC. The results will be shared with other Military Health System (MHS) and Veterans Health Administration (VHA) pain management centers so that active duty Service members and veterans across United States may benefit from a treatment approach that is tailored to their individual characteristics. It is anticipated that the knowledge gained through this research will be applicable to family members of Service members and veterans and will ultimately lead to expansion of TRICARE benefits to include CIM therapies.

Potential Clinical Applications, Benefits, and Risks. This research will assist providers in determining when to refer their patients with neuromusculoskeletal pain for SRC and/or CIM therapies prior to FR. It will assist IPMCs in developing treatment plans tailored to the needs of each patient. Service members and veterans will benefit by being referred for these approaches when appropriate during the course of disabling chronic pain conditions. Ultimately, it is hoped that decision tools can be imbedded in the electronic medical record to guide health care providers to consider referral for these therapies in patients who may benefit. This study will advance our ability to effectively tailor therapies for rehabilitation from neuromusculoskeletal pain for different patients to yield the greatest benefit in physical function and quality of life. The risks of these interventions are minimal; Service members may experience general muscle soreness for the first week or so of increased physical activity, but this typically resolves.

Projected Timeline. This research will determine the optimal combination, sequence, and duration of therapies. It is expected that some active duty Service members could see improvements in function and quality of life within three weeks, but others may require up to six weeks to experience meaningful improvement.

Benefit to Military Personnel. This research will benefit Service members experiencing pain due to neuromusculoskeletal injury. It will identify ways to direct them to the therapies most likely to yield meaningful improvements in function and quality of life, and thus facilitate their return to duty. The recommendations from this study will be shared with pain management centers throughout the DoD, VHA; and, we hope, eventually to TRICARE members.

ELIGIBILITY:
Inclusion Criteria:

* Active duty service members
* Neuromusculoskeletal or neuropathic pain ≥ 3-months duration
* Pain of sufficient severity to bring about dysfunction in daily social, vocational, and/or interpersonal activities

Exclusion Criteria:

* Major surgeries within past 6 months or planned within next 6 months
* Unstable psychological disorders
* Active substance use disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Pain Intensity | 3 months
  Pain Intensity 10-pt Numeric Rating Scale
Change from Baseline Pain Impact | 3 months
  Aggregate score calculated from Defense and Veterans Pain Rating Scale (DVPRS)

SECONDARY OUTCOMES:
Depression | baseline, 3 weeks, 6 weeks, 9 weeks, 3 months, 6 months
  Patient Reported Outcome Measurement Information System
Anxiety | baseline, 3 weeks, 6 weeks, 9 weeks, 3 months, 6 months
  Patient Reported Outcome Measurement Information System
Emotional Distress - Anger | baseline, 3 weeks, 6 weeks, 9 weeks, 3 months, 6 months
  Patient Reported Outcome Measurement Information System
Sleep Disturbance | baseline, 3 weeks, 6 weeks, 9 weeks, 3 months, 6 months
  Patient Reported Outcome Measurement Information System
Fatigue | baseline, 3 weeks, 6 weeks, 9 weeks, 3 months, 6 months
  Patient Reported Outcome Measurement Information System
PTSD | baseline, 3 weeks, 6 weeks, 9 weeks, 3 months, 6 months
  Primary Care PTSD Screen
Patient Activation Measure | baseline, 3 weeks, 6 weeks, 9 weeks, 3 months, 6 months
  A 22-item survey that addresses four stages of patient activation: (1) believing the patient role is important, (2) having the confidence and knowledge necessary to take action, (3) actually taking action to maintain and improve one's health, and (4) staying the course even under stress. Patients are asked to agree or not to agree with each of the 22 items.
Drug Use | baseline, 3 weeks, 6 weeks, 9 weeks, 3 months, 6 months
  Drug Use Questionnaire
Pain Catastrophizing | baseline, 3 weeks, 6 weeks, 9 weeks, 3 months, 6 months
  Pain Catastrophizing Scale
Kinesiophobia | baseline, 3 weeks, 6 weeks, 9 weeks, 3 months, 6 months
  Tampa Scale for Kinesiophobia
Pain Self-Efficacy | baseline, 3 weeks, 6 weeks, 9 weeks, 3 months, 6 months
  Pain Self Efficacy Questionnaire
Chronic Pain Acceptance | baseline, 3 weeks, 6 weeks, 9 weeks, 3 months, 6 months
  Chronic Pain Acceptance Questionnaire
Functional Capacity | baseline, 3 weeks, 6 weeks, 9 weeks, 3 months, 6 months
  Roland-Morris Disability Questionnaire and Canadian Occupational Performance Measure
Opioid Utilization | baseline, 3 weeks, 6 weeks, 9 weeks, 3 months, 6 months
  Opioid Utilization Screener
Cortisol | baseline, 6 weeks
  Salivary Cortisol
Oxidative Stress | baseline, 6 weeks
  Urine Sample
Genomic DNA | baseline
  Buccal Sample
Army Physical Fitness Test (APFT) | baseline, 6 weeks, 3 months, 6 months
  Passing scores of 60 on all 3 components (push-ups, sit-ups, 2-mile run) of the APFT will be operationalized as "force-readiness".

CONTACTS AND LOCATIONS:
Overall Officials: Ardith Z Doorenbos, RN, PhD, Principal Investigator — University of Washington
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

REFERENCES:
- [Derived] Shimada S, Ledesma S, Flynn DM, Tintle N, Ransom JC, McQuinn HM, Snow TJ, Ieronimakis N, Wi D, Burke LA, Steffen AD, Doorenbos AZ. Evaluating Sex Differences in Biomarkers of Chronic Pain Among Active-Duty Personnel: An Exploratory Analysis of a Pragmatic Clinical Trial With a SMART Design. Biol Res Nurs. 2026 Feb 3:10998004261423210. doi: 10.1177/10998004261423210. Online ahead of print. PMID 41631713
- [Derived] Wi D, Flynn DM, Park C, Ransom JC, McQuinn HM, Snow TJ, Burke LA, Steffen AD, Shimada S, Doorenbos AZ. Dynamic Interactions in Chronic Pain-Related Outcomes: A Secondary Data Analysis of a Pragmatic Clinical Trial With Sequential, Multiple Assignment, Randomized Trial Design. Mil Med. 2025 Nov 1;190(11-12):e2382-e2390. doi: 10.1093/milmed/usaf225. PMID 40440185
- [Derived] Flynn DM, Ransom JC, Steffen AD, Orr KP, McQuinn HM, Snow TJ, Burke LA, Wi D, Doorenbos AZ. Complementary, integrative, and standard rehabilitative therapies in a military population with chronic predominantly musculoskeletal pain: a pragmatic clinical trial with SMART design. Pain. 2025 Jun 1;166(6):1343-1353. doi: 10.1097/j.pain.0000000000003462. Epub 2024 Nov 8. PMID 39560398